CLINICAL TRIAL: NCT07300280
Title: A Clinical Study to Evaluate the Relative Bioavailability of an FDC Tablet Containing Enlicitide and Rosuvastatin, Compared to Enlicitide and Rosuvastatin Administered Concomitantly as Single Entities, in Healthy Adult Participants
Brief Title: A Clinical Trial of Enlicitide and Rosuvastatin in Healthy Adults (MK-0616-039)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616A-039
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enclidite + Rosuvastatin (Experimental): Participants will receive a single dose of enlicitide tablet coadministered with a single dose of rosuvastatin tablet
  Interventions: Drug: Enlicitide; Drug: Rosuvastatin
- MK-0616A (Experimental): Participants will receive a single dose of MK-0616A
  Interventions: Drug: MK-0616A

INTERVENTIONS:
Drug: MK-0616A — Enlicitide/rosuvastatin fixed dose combination (FDC) oral tablet
  Other Names: enlicitide/rosuvastatin calcium
  Arms: MK-0616A
Drug: Enlicitide — Oral tablet
  Other Names: MK-0616
  Arms: Enclidite + Rosuvastatin
Drug: Rosuvastatin — Oral tablet
  Arms: Enclidite + Rosuvastatin

SUMMARY:
This goal of this trial is to learn about two medicines, enlicitide and rosuvastatin, in healthy people. Researchers will compare the amounts of enlicitide and rosuvastatin in a person's body over time, when they are given as separate medicines and when they are combined into one tablet.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Is medically healthy with no clinically significant medical history
* Is a non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to study entry

Exclusion Criteria:

* Is unable to refrain from or anticipates the use of any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to study entry
* Is a female participant of childbearing potential

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Enlicitide | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the AUC0-inf of enlicitide in plasma
AUC0-Inf of Rosuvastatin | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the AUC0-inf of rosuvastatin in plasma
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Enlicitde | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the AUC0-last of enlicitide in plasma
AUC0-Last of Rosuvastatin | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the AUC0-last of rosuvastatin in plasma
Maximum Plasma Concentration (Cmax) of Enlicitide | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the cmax of enlicitide in plasma
Cmax of Rosuvastatin | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the cmax of rosuvastatin in plasma
Time to Maximum Plasma Concentration (Tmax) of Enlicitide | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the tmax of enlicitide in plasma
Tmax of Rosuvastatin | Pre dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the tmax of rosuvastatin in plasma

SECONDARY OUTCOMES:
Number of Participants who Experience an Adverse Event (AE) | Up to approximately 9 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 8 days after first dose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com